CLINICAL TRIAL: NCT06659432
Title: Relationship Between Sensory Profile and Academic Achievement in University Students
Brief Title: Sensory Profile and Academic Achievement in Students
Status: Active, not recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Associate Professor, Gazi University
Other Study IDs: 87881925
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: University Students
Keywords: Sensation disorders; Students; Academic success
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Senses are fundamental to the neurological system, enabling individuals to perceive their bodies and interact with their surroundings. While the five primary senses-vision, smell, hearing, taste, and touch-are well known, humans also possess three "hidden" senses: the vestibular sense (movement and gravity), proprioception (body position), and interoception (internal organs). Sensory integration, as defined by Dr. Jean Ayres, is the process of receiving, processing, and generating motor responses to sensory input, which influences learning, behaviors, and personality traits. Dr. Winnie Dunn's "Four Quadrant Model of Sensory Processing" further explores how individuals respond to sensory stimuli based on their neurological thresholds and behavioral responses. The model includes four quadrants: low registration, sensation seeking, sensory sensitivity, and sensation avoiding, each of which affects behaviors in daily life, including educational settings. For example, a student with low registration may need more stimuli to focus, while a sensation-avoiding student may prefer quieter environments. Research shows that sensory processing influences academic achievement, yet studies on this relationship in young adults are limited. This study aims to assess how sensory processing impacts academic success among university students.

DETAILED DESCRIPTION:
The nervous system in our body consists of various sensory systems, such as the visual, gustatory, olfactory, auditory, tactile, and vestibular senses, which enable us to receive and process stimuli from the environment. Ayres and Robbins defined sensory processing as a neurological process that organizes the sensory input received from the body and environment, allowing us to use the body effectively in our surroundings. This process is natural for humans and continues throughout life, without being limited to a specific age. When sensory processing issues arise, difficulties in adapting to the environment and using the body effectively can occur, leading to confusing social behaviors. Additionally, it becomes challenging to understand the atmosphere of the environment and the words and behaviors of others, resulting in slow responses to stimuli and difficulties in social activities and interpersonal relationships. In adults, challenges in sensory processing abilities can negatively affect attention, lead to inappropriate sensory regulation and defence, cause maladaptive behaviors, and impact academic success.

Just as work is a significant area of life for professionals, learning is a major aspect of life for university students. The university years are a critical period in Erikson's developmental stages for discovering and establishing identity. For university students, learning is a choice for continuous growth and self-regulation, adding meaning to life. Learning at university differs from secondary and high school education; the role of the learner shifts from passive to active, requiring them to manage their own learning. This creates significant differences in the amount and depth of knowledge acquired, depending on the learner's abilities. Today, with the overwhelming amount of available information, it is impossible to convey all necessary knowledge in a classroom setting. Students must develop the ability to independently evaluate and select the information they need. University learning offers greater independence and autonomy compared to other educational periods, and learning strategies that enhance efficiency play an important role in academic success.

Academic achievement is a comprehensive concept that reflects the extent to which individuals attain their educational goals. Various studies have identified internal and external factors that affect academic success. In recent years, sensory processing issues have been added to these factors, drawing the attention of researchers. According to Dunn's model, students with different sensory processing profiles may exhibit various behaviors in the learning environment: A "low registration" student may struggle to focus during class when not exposed to adequate stimulation and may prefer taking notes over actively following the lesson. A "sensation seeking" student may require continuous stimuli to stay focused and might satisfy this need by biting a pen or fidgeting. A student with "sensory sensitivity" might be disturbed by complex presentations in the classroom and have difficulty concentrating. A "sensation avoiding" student, on the other hand, may be bothered by classroom noise and the presence of other students and may choose to sit at the front of the class to concentrate better. These behaviors illustrate how sensory processing affects academic success. Despite its significance, research exploring the connection between sensory processing and academic performance in young adults remains limited. Therefore, this study aimed to evaluate the relationship between sensory processing and academic achievement in university students.

ELIGIBILITY:
Inclusion Criteria:

* To be a student in the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Gazi University

Exclusion Criteria:

* Students who declined to participate
* Students who incomplete the survey forms

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: University Students
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Adolescent/Adult Sensory Profile Questionnaire | 1 day
  The AASP, a 60-item self-report questionnaire, was used to evaluate participants' sensory processing by assessing their responses to various sensory stimuli, including taste/smell, movement, visual, touch, auditory processing, and activity level. Evaluation was conducted using a five-point Likert scale. Higher scores reflect a greater manifestation of specific sensory processing traits. The items in each section were combined into four quadrants to characterize experience and behavior. These quadrants are grouped as "low registration," "sensation seeking," "sensory sensitivity," and "sensation avoidance" . We used the Turkish version of the AASP in present study.

SECONDARY OUTCOMES:
Academic Achievement | Two months
  Academic success scores of university students are examined.

CONTACTS AND LOCATIONS:
Overall Officials: Muserrefe Nur Keles, PhD, Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided